CLINICAL TRIAL: NCT05358639
Title: A Phase I Trial of the Combination of Olaparib and Navitoclax in Women with High Grade Serous Epithelial Ovarian Cancer and Triple Negative Breast Cancer
Brief Title: Combination of Olaparib and Navitoclax in Women with HGSC and TNBC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Exactis Innovation (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exactis-03
Record Dates: First submitted 2022-03-22; First posted 2022-05-03 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: High Grade Serous Carcinoma; Triple Negative Breast Cancer; Ovarian Cancer
Keywords: BRCA1 Mutation; BRCA2 Mutation; PALB2 Gene Mutation; Olaparib; Navitoclax; Bcl-2; Bcl-xL; Bax; Mcl-1; Bcl-W; Bak; Bok; Bid; Bim; Bad; Bik; Noxa; Puma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Ovarian Neoplasms | interventions — olaparib; navitoclax

STUDY DESIGN:
Intervention Model Description: The trial is designed as an open-label multi-center Phase I interventional and translational study. It will identify the dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) and RP2D of olaparib combined with navitoclax for study in Phase II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single (Experimental): Olaparib tablet will be administered alone for 14 days at a starting dose of 200 mg twice daily (bid). Subsequently olaparib will be administered continuously over 28 days at a fixed dose and the dose of navitoclax will be escalated. Navitoclax will be administered daily. The initial dose of olaparib 200 mg has been selected after considering the single agent Phase I/II dose based and on ongoing combination studies on expected toxicity and evidence for reduced PARP inhibition
  Interventions: Drug: Olaparib tablet; Drug: Navitoclax

INTERVENTIONS:
Drug: Olaparib tablet — Olaparib tablet will be administered alone for 14 days at a starting dose of 200 mg twice daily. Subsequently olaparib will be administered continuously over 28 days at a fixed dose and the dose of navitoclax will be escalated.
  Other Names: Lynparza
Drug: Navitoclax — For navitoclax, a lead-in of 7 days at 150 mg PO will be used prior to dose escalation. The DLT period for dose levels above DL 3 will include the 14-day olaparib alone lead-in, the 7 days combination with navitoclax at 150 mg and the first 28 day cycle of the combination of olaparib and navitoclax cycle at the full dose level dosing (49 days).
  Other Names: ABT-263

SUMMARY:
The purpose of this Phase I study is to determine if the PARP inhibitor olaparib can be safely combined with navitoclax, an inhibitor of Bcl-2/Bcl-XL, in women with TNBC who have somatic or germline mutations in breast cancer gene one (BRCA1) and breast cancer gene two (BRCA2) BRCA1/2 or PALB2 and in women with recurrent HGSC who have progressed greater than 6 months since their last platinum containing chemotherapy. The trial is designed as an open- label multi-center Phase I interventional and translational study. It will identify the dose-limiting toxicities (DLTs), maximum tolerated dose (MTD) and RP2D of olaparib combined with navitoclax for study in Phase II. There is a plan for a follow on Phase II study depending on the results obtained during this Phase I trial.The rationale for this study is that for a subset of patients, olaparib, will increase tumor cell survival dependence on inhibition of cell death by Bcl 2/Bcl- XL. Thus, navitoclax will augment apoptosis induced by PARP inhibition with olaparib.

DETAILED DESCRIPTION:
In this trial, olaparib will be delivered alone for 14 days with the hypothesis that priming of the apoptotic machinery will be required prior to introduction of the senolytic agent (navitoclax). To date navitoclax and olaparib have not been combined in the clinic. The Phase I study will therefore be conducted to define the recommended Phase II dose (RP2D). A plan for a future Phase II study will depend on the results obtained during this Phase I trial. Based on the potential for overlapping toxicity (particularly hematologic toxicity) an interrupted dosing schedule will be used for the navitoclax. Based on preclinical studies it is believed that intermittent delivery of the senolytic agent is in line with the proposed mechanism of action. Subsequently the dose of navitoclax will be escalated with a fixed dose of olaparib in 28-day cycles.

ELIGIBILITY:
Inclusion

* Histologically confirmed:

  * Recurrent metastatic HGSC of ovarian, peritoneal or fallopian tube origin with radiological progression greater than 6 months from last platinum based therapy.
  * Metastatic TNBC: tumors that are known to have deleterious somatic or germline mutations in BRCA1, BRCA2, or PALB2.

    * Age ≥ 18 years of age.
    * ECOG Performance Status of 0, 1 or 2 within 7 days prior to registration (Appendix 4).
    * No more than two (2) prior lines of treatment for TNBC.
    * No limit on the number of prior lines for HGSC.
    * Prior maintenance or treatment with PARP inhibitor is allowed provided progression did not occur on or within 6 months of discontinuing the drug. Patients must be considered able to tolerate olaparib as per dosing regimen in this study.
    * Patients must be able to swallow and retain oral medications and without gastrointestinal illnesses that would preclude absorption.
    * Patients must be able and willing to undergo study related procedures (biopsies pre and on treatment) and to provide archival tissue, if available.
    * Patients must have a life expectancy ≥16 weeks.
    * Patients must have adequate organ and marrow function measured within 28 days prior to administration of study drug
* Patients must have measurable disease as defined by RECIST 1.1. Progressive irradiated lesions considered but would require an additional out of field measurable lesion.

  * Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

Exclusion

* Prior chemotherapy, endocrine therapy, radiotherapy, or investigational agents within 30 days prior to first dose of investigational products (IPs).
* Due to the expected dose-limiting toxicity of thrombocytopenia, the following concomitant medications are not allowed within 14 days of the olaparib lead-in period: Warfarin, clopidogrel (plavix), ibuprofen, tirofiban (aggrastat), and other anticoagulants drugs including low molecular weight heparin, or herbal supplements that affect platelet function are excluded. Caution should be exercised when dosing Navitoclax concurrently with CYP2C8 and CYP2C9 substrates.
* Due to the known effects of navitoclax on platelet counts, patients with active bleeding or thrombocytopenia-associated bleeding within 1 year, active peptic ulcer disease or potentially hemorrhagic esophagitis or gastritis, a requirement for concurrent therapeutic anticoagulants, or a history of immune thrombocytopenic purpura, autoimmune hemolytic anemia, or refractoriness to platelet transfusions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
To define a dose and schedule of navitoclax (Recommended Phase II Dose, RP2D) that can be combined safely with Olaparib in women with metastatic recurrent high grade serous ovarian cancer (HGSC) and triple negative breast cancer (TNBC) for further study | 2 years
  The RP2D will be determined based on an evaluation of multiple endpoints, which will include the DLT( dose limiting toxicity) rate.

SECONDARY OUTCOMES:
Cmax: the maximum drug concentration. | 2 years
  The maximum drug concentration will be measured in blood samples as part of the PK profile of olaparib and navitoclax when given in combination.
Tmax: time to reach the maximum drug concentration. | 2 years
  The time to reach maximum drug concentration will be measured in blood samples as part of the PK profile of olaparib and navitoclax when given in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Helen MacKay, MD, Principal Investigator — Sunnybrook Cancer Centre
Locations (3):
- Canada (3):
  - Sunnybrook Research Institute/Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No